CLINICAL TRIAL: NCT00131820
Title: Introduction of the Vi Polysaccharide Typhoid Vaccine in Hue City, Central Vietnam. An Evaluation of Feasibility, Public Acceptability, Effectiveness and Cost-Effectiveness in Students
Brief Title: Introduction of the Vi Polysaccharide Typhoid Vaccine in Hue City, Central Vietnam
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: National Institute of Hygiene and Epidemiology, Vietnam (Other); Hue Preventive Medicine Center, Vietnam (Unknown); Wellcome Trust (Other); University of Western Ontario, Canada (Other); GlaxoSmithKline (Industry)
Responsible Party: Mr. Leon Ochiai, International Vaccine Institute
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: T-14
Record Dates: First submitted 2005-08-18; First posted 2005-08-19 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-03

CONDITIONS: Typhoid; Paratyphoid Fever
Keywords: Salmonella; typhoid vaccine; enteric fever; socioeconomic costs
MeSH Terms: conditions — Typhoid Fever; Paratyphoid Fever | interventions — Vi polysaccharide vaccine, typhoid; Hepatitis A Vaccines

INTERVENTIONS:
Biological: Typhoid Vi vaccine
Biological: Hepatitis A (control)

SUMMARY:
This study is part of International Vaccine Institutes (IVI)'s typhoid Vi demonstration project that aims to accelerate the rational introduction of Vi vaccines in typhoid endemic countries. The primary objectives of the study are to evaluate the logistic feasibility of a mass typhoid fever immunization campaign program targeting school age children in Hue City, Vietnam and to assess the knowledge, attitudes, beliefs, and practices of parents and healthcare providers in Hue City regarding typhoid fever prevention and treatment.

DETAILED DESCRIPTION:
Typhoid fever is a major cause of morbidity worldwide. The disease predominantly affects school-aged children, is more prevalent in urban areas, may last for several weeks and can lead to serious complications. Management of this disease is further complicated by the emergence of multi-drug resistant strains. Vaccination of high risk populations is considered the most promising strategy for the control of typhoid fever. The Vi polysaccharide vaccine has been targeted for accelerated introduction into public health programs due to the following reasons: it has been shown to have consistent efficacy results even in areas of high typhoid incidence, is given as a single dose, lacks patent protection and requires less strict cold chain requirements. A cluster-randomized trial involving the Vi polysaccharide vaccine and an active control (Hepatitis A) was designed to determine the logistic feasibility of providing Vi vaccine under actual programmatic conditions among school students in Hue City. The vaccines used in this study are internationally produced and locally licensed.

Secondary objectives of this trial are:

* To estimate the cost-effectiveness (cost of illness, willingness to pay, vaccine delivery costs, private vaccine costs, etc) of Vi vaccination
* To determine the effectiveness of the Vi polysaccharide vaccine following routine administration of a 1-dose schedule to school students (aged >=6 years)
* To determine the safety and immunogenicity of the Vi vaccine
* To study typhoid risk factors among students

A nested, prospective matched case-control study is included in the trial in order to study typhoid risk factors among children in Hue City.

ELIGIBILITY:
Inclusion Criteria:

* Local students whose parents/guardians provide written consent to receive Vi vaccine
* Attending any of the 66 registered schools in Hue
* Registered in the project census
* Lives in Hue City

Exclusion Criteria:

* Fever (>37.5 degrees Celsius, axillary)
* Pregnancy
* Lactating

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100742
Dates: Start 2001-12; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Logistic feasibility of mass typhoid immunization campaign
Knowledge attitudes, beliefs and practices of parents and health care providers on typhoid fever prevention and treatment

SECONDARY OUTCOMES:
Cost-effectiveness of vaccine
Vaccine effectiveness
Adverse events
Typhoid risk factors

CONTACTS AND LOCATIONS:
Overall Officials: Canh G Do, MD, Principal Investigator — National Institute of Hygiene and Epidemiology, Vietnam
Locations (1):
- National Institute of Hygiene and Epidemiology, Hanoi, Vietnam

REFERENCES:
- [Background] Acosta CJ, Galindo CM, Ochiai RL, Danovaro-Holliday MC, Page AL, Thiem VD, Park JK, Park E, Koo H, Wang XY, Abu-Elyazeed R, Ali M, Albert MJ, Ivanoff B, Pang T, Xu ZY, Clemens JD. The role of epidemiology in the introduction of vi polysaccharide typhoid fever vaccines in Asia. J Health Popul Nutr. 2004 Sep;22(3):240-5. PMID 15609776